CLINICAL TRIAL: NCT06906276
Title: Walking and Thinking - Brain Activity During Complex Walking in Atypical Parkinsonian Syndromes
Brief Title: Brain Activity During Complex Walking in People With Atypical Parkinsonian Syndromes
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Erika Franzén, Professor Erika Franzén, RPT, PhD, Karolinska Institutet
Other Study IDs: 4-2452/2024; 2020-03059 (Other: other Study ID)
Record Dates: First submitted 2025-03-12; First posted 2025-04-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-03

CONDITIONS: Gait Disorders, Neurologic; Atypical Parkinson Disease; fNIRS; Aging
MeSH Terms: conditions — Gait Disorders, Neurologic; Parkinson Disease, Familial, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Atypical Parkinsonian syndromes: -People with either Progressive supranuclear palsy or Multiple system atrophy
  Interventions: Other: Assessment of brain activity with fNIRS and behavioural assessments (motor, motor-cognitive and cognitive) during three complex walking conditions.

INTERVENTIONS:
Other: Assessment of brain activity with fNIRS and behavioural assessments (motor, motor-cognitive and cognitive) during three complex walking conditions. — Dual-task walking with the auditory stroop task. Navigational walking - a course consisting of a distribution of 45 and 90 degrees turns to the left and right Navigational and dual-task walking (condition 1 and 2 together)

SUMMARY:
Every-day life means being part of a complex environment and performing complex tasks that usually involve a combination of motor and cognitive skills. However, the process of aging or the sequelae of neurological diseases such as atypical Parkinson's disease (APD) compromises motor-cognitive interaction necessary for an independent lifestyle. While motor-cognitive performance has been identified as an important goal for sustained health across different clinical populations, little is known about underlying brain function leading to these difficulties and how to best target these motor-cognitive difficulties in the context of rehabilitation and exercise interventions.

The challenge of improving treatments of motor-cognitive difficulties (such as dual-tasking and navigation) is daunting, and an important step is arriving at a method that accurately portrays these impairments in an ecologically valid state. The investigators aim therefore to explore brain function during complex walking in healthy and APD by investigating the effects of age and neurological disease on motor-cognitive performance and its neural correlates during three conditions of complex walking (dual-task walking, navigation and a combination of both) using non-invasive measures of brain activity (functional near infrared spectrometry, fNIRS) and advanced gait analysis in real time in older healthy adults and people with APD.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of PSP according to Movement Disorder Society (MDS) (2017) or
* MSA according to MDS criteria (2022)
* the ability to walk with or without a mobility device for ≤5 minutes continuously

Exclusion Criteria:

* cognitive difficulties affecting the ability to understand and/or follow verbal/written - instructions
* severe freezing of gait
* Severe hearing or visual impairments that affect participation in the assessments
* Other neurological diseases
* Other diseases that can affect gait or balance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are studying complex walking in different populations, such as people with Multiple Sclerosis, healthy young adults, healthy elderly, and elderly with Parkinson's disease. We have during 2022 completed data collection (ClinicalTrials.gov ID: NCT05218213) of healthy young adults, healthy elderly, and elderly with Parkinson's disease. In 2024, we completed data collection in people with Multiple Sclerosis (NCT05787704).
  Hence, this registration concerns the atypical parkinsonism cohort.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional near infrared spectrometry (fNIRS) | Baseline
  The measurement of changes in concentration of HbO and HHb in the prefrontal cortex will be assessed using a NIRSPORT 2 (NIRx Medizintechnik, Berlin, Germany) device.
Gait performance during all conditions | Baseline
  Gait variables such as stride time and/or velocity will be analyzed with the APDM mobility system.
Dual-task performance-reaction time | Baseline
  Cognitive performance of the dual task will be assessed as errors in the response to the Auditory Stroop task.

SECONDARY OUTCOMES:
Resting-state functional near infrared spectrometry (rsfNIRS) | Baseline
  The measurement of changes in concentration of HbO and HHb in the whole cortex will be assessed using a NIRSPORT 2 (NIRx Medizintechnik, Berlin, Germany) device during 2x 10min of rest, while seated in a comfortable chair.
Cognitive function- composite score | Baseline
  The cognitive test battery comprised the following tests: The Color-Word Interference Test (CWIT), Verbal Fluency, Trail Making Test (TMT), Ray Auditory Verbal Learning Test (RAVLT), and Symbol Digit Modalities Test (SDMT). Cognitive function will be assessed as a composite measure of these tests together.
Cognitive function - verbal fluency | Baseline
  Verbal function, initiation & task-set switching with the Verbal Fluency test from D-KEFS (Delis-Kaplan Executive Function System).
Cognitive function - Attention and psychomotor processing speed | Baseline
  Attention and psychomotor processing speed will be assessed with the Trail Making Test (TMT) from D-KEFS (Delis-Kaplan Executive Function System).
Cognitive function - Episodic memory | Baseline
  Episodic memory will be assessed with the Ray Auditory Verbal Learning Test (RAVLT).
Cognitive function - Inhibition & task-set switching | Baseline
  Inhibition & task-set switching with the Color-Word Interference Test (CWIT) from D-KEFS (Delis-Kaplan Executive Function System)
Self-reported level of physical activity | Baseline
  Assessed with the Frändin-Grimby Scale (score 1-6, higher score=better)
Physical activity | Baseline
  Assessed with accelerometers (Actigraph GT3X+) for seven consecutive days after the clinical visit
Motor function/disease severity | Baseline
  Assessed with the movement Disorders Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Higher scores = worse/more symptoms
Balance performance | Baseline
  Assessed with the Mini-BESTest (Balance Evaluation Systems test), 0-28p,
Anxiety and depression | Baseline
  Assessed with Hospital Anxiety and Depression Scale (HADS), 0-24 on the depression and anxiety part respectively. Lower score=better
Walking ability | Baseline
  Self-assessed walking ability with the WALK-12G.
Dual-task performance -errors | Baseline
  Cognitive performance of the dual task will be assessed as the reaction time to respond during the Auditory Stroop
Disability | Baseline
  WHO Disability Assessment Schedule (WHODAS) version 2.0, 12 self-assessed questions (12 to 60) more points=worse

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Albrecht, PhD, Principal Investigator — Karolinska Institutet; Erika Franzén, Prof,, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and EU personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient, provided that the recipient has an approved ethics application.
Supporting Information: SAP, Analytic Code
Time Frame: We plan to share this when applicable on OSF
Access Criteria: The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and EU personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient.
URL: https://osf.io/btnz6/?view_only=5de87008a47f4cc0b839906accdb2da5